CLINICAL TRIAL: NCT07121595
Title: PRECEDENT: Pilot Phase II Study of Personalized Radiation to the Contralateral Neck Directed by Sentinel Node Evaluation in Lateralized Oral Cavity Squamous Cell Carcinoma
Brief Title: Personalized Neck Radiation Therapy Directed by Sentinel Lymph Node Biopsy for the Treatment of Oral Cavity Squamous Cell Carcinoma, PRECEDENT Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2023.022; NCI-2025-01191 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00258370 (Other: University of Michigan Rogel Cancer Center)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Oral Cavity Squamous Cell Carcinoma; Stage I Lip and Oral Cavity Cancer AJCC v8; Stage II Lip and Oral Cavity Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage IVA Lip and Oral Cavity Cancer AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Mouth Neoplasms | interventions — Specimen Handling; Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Paclitaxel; Taxes; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation; Sentinel Lymph Node Biopsy; X-Rays; Photons; technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (SLN mapping, SLNB, RT, chemotherapy) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Modified Barium Swallow; Drug: Paclitaxel; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy; Procedure: Sentinel Lymph Node Biopsy; Procedure: Single Photon Emission Computed Tomography; Radiation: Technetium Tc 99m-labeled Tilmanocept; Other: Technetium Tc-99m Sulfur Colloid

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT and/or SPECT-CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Modified Barium Swallow — Undergo video fluoroscopic swallow study
  Other Names: MBS; VFSS; Videofluoroscopic Swallowing Study
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Procedure: Positron Emission Tomography — Undergo PET-CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Procedure: Sentinel Lymph Node Biopsy — Undergo SLNB
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT-CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Technetium Tc 99m-labeled Tilmanocept — Given via injection
  Other Names: 99mTc-Diethylenetriamine Pentaacetic Acid-Mannosyl-Dextran; 99mTc-DTPA-Mannosyl-Dextran; Lymphoseek; Tc99m Tilmanocept; TECHNETIUM TC-99M TILMANOCEPT
Other: Technetium Tc-99m Sulfur Colloid — Given via injection
  Other Names: Tc 99m Sulfur Colloid; Tc-99m SC; Technetium Tc 99m Sulfur Colloid

SUMMARY:
This phase II trial studies how well personalized neck radiation therapy directed by sentinel lymph node biopsy (SLNB) works in treating patients with oral cavity squamous cell carcinoma (OCSCC). SLNB can be performed as part of standard care for OCSCC. During SLNB, a radiotracer is injected around the tumor. The lymph nodes are then biopsied and tested to see if the tracer injected into the tumor traveled to and is present in the sentinel lymph nodes (SLNs). Results of the SLNB are used to determine whether lymph nodes should be removed in both sides of the neck or just on the same side as the primary tumor. Standard treatment then involves radiation therapy to both sides of the neck, regardless of SLNB results. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. Studies have shown only a small number of patients develop a return of the cancer (recurrence) in the opposite side of the neck after radiation therapy. In addition, radiation therapy can negatively impact patient outcomes like saliva production, speech and swallow function, increased risk of radiation induced cancers, and chronic pain. Standard of care SLNBs may be effective in determining whether radiation therapy only needs to be administered to one side of the neck or both sides. This may help spare tissue on the opposite side of the neck from receiving radiation if there is no indication of lymph node involvement there.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have biopsy-proven squamous cell carcinoma of the oral cavity
* Clinical stage cT1-4a N0-2b M0 within 42 days of study enrollment based on the following work-up:

  * History and physical examination within 42 days of study enrollment; must include documentation of lateralized primary tumor site
  * Cross-sectional imaging of the head and neck within 42 days of study enrollment
  * Cross-sectional imaging of the chest within 42 days of study enrollment
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2 within 42 days of study enrollment
* Age > 18
* Recommended treatment plan is surgical resection with ipsilateral neck dissection and SPECT-CT-guided sentinel node biopsy. Flap reconstruction is allowed
* Patient is willing and able to provide informed consent. Patient provides study-specific informed consent prior to study entry
* Women of childbearing potential and male participants must agree to use medically effect means of birth control throughout their participation in the treatment phase of the study

Exclusion Criteria:

* Evidence of distant metastatic disease based on clinical or radiologic evaluation
* Evidence of contralateral neck disease on staging imaging
* Prior non-head and neck invasive malignancy (except non-melanomatous skin cancer, including effectively treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or cervix) unless disease free for ≥ 2 years
* Diagnosis of head and neck squamous cell carcinoma (SCC) in the oropharynx, nasopharynx, hypopharynx, and larynx
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowed. Prior immunotherapy for the study cancer is allowed.
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Patient with severe, active co-morbidity that would preclude an elective or completion neck dissection
* Pregnant and breast-feeding patients
* Excisional biopsy for study cancer
* Prior surgery involving the lateral neck, including neck dissection or gross injury to the neck that would preclude surgical dissection for this trial. Prior thyroid and central neck surgery is permissible; incisional biopsy is permitted
* Underlying or documented history of hematologic malignancy (e.g., chronic lymphocytic leukemia [CLL]) or other active disease capable of causing lymphadenopathy (sarcoidosis or untreated mycobacterial infection)
* Actively receiving systemic cytotoxic chemotherapy, immunosuppressive, anti-monocyte or immunomodulatory therapy
* Currently participating in another investigational therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Contralateral regional control rate | From completion of definitive treatment to neck recurrence date, death date or date of last contact, assessed at 1 year from completion of definitive treatment
  Contralateral regional control rate is defined as the proportion of evaluable subjects free of contralateral neck recurrence at 1 year from completion of definitive treatment. Regional Recurrence is defined as biopsy-proven cancer within the ipsilateral or contralateral neck at any time point after initial surgical resection. When biopsy is not feasible, evidence of recurrence by imaging suffices only with documented attestation at tumor board that the imaging is clinically diagnostic of regional recurrence. Cumulative incidence function estimate with 90% confidence interval (CI) for follow-up after 1 year.

SECONDARY OUTCOMES:
Change in neck function | Baseline up to 1 year from completion of definitive treatment
  Will be assessed using five number summary* (minimum [min], first quartile [Q1], median, third quartile [Q3], maximum [max]) of Neck Dissection Impairment Index summary scores.
Change in oral and oropharyngeal dryness | Baseline up to 3 months from completion of definitive treatment
  Will be assessed using five number summary* (min, Q1, median, Q3, max) of summary score on the Xerostomia questionnaire.
Change in quality of life | Baseline up to 3 months from completion of definitive treatment
  Will be assessed using five number summary* (min, Q1, median, Q3, max) of summary score on the University of Washington Quality of Life Survey, a 15-item survey evaluating quality of life metrics focused on speech, eating, saliva, taste, phlegm, employment, recreation, activity, disfigurement, and pain.
Recurrence free survival | 1 year from completion of definitive treatment
  Will assess # evaluable, # events and # censored at 1 year from completion of definitive treatment, as well as Kaplan-Meier (KM) estimate with 95% CI.
Overall survival | 1 year from completion of definitive treatment
  Will assess # evaluable, # events and # censored at 1 year from completion of definitive treatment, as well as KM estimate with 95% CI.
Disease-specific survival | 1 year from completion of definitive treatment
  Will assess # evaluable, # events and # censored at 1 year from completion of definitive treatment, as well as KM estimate with 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Shah, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States